CLINICAL TRIAL: NCT06692413
Title: Withings Devices Follow-up Study - Hypertension
Status: Enrolling by invitation | Type: Observational
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: WIQUEST-HTA
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Withings device users: Active Withings device users having at least 2 years of device data
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Users who consent to the study will receive a questionnaire every 3 months

SUMMARY:
The primary objective is to evaluate the accuracy to predict uncontrolled hypertension with Withings device data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who are 21 years of age or older,
* Participant living in the United States,
* Participant with data recorded in WITHINGS database,
* Active WITHINGS device users having at least 2 years of data,
* Subject able to read, understand, and provide written informed consent,
* Subject willing and able to participate in the study procedures as described in the consent form,
* Subject able to communicate effectively with and willing to follow instructions from the study staff.

Exclusion Criteria:

* Minors under 21 years old,
* Subject who refused to participate in the study,
* Subject who did not reply to the questionnaire,
* Subject who objected to the processing of his or her data after the start of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population meeting the inclusion criteria will all live in the US, regular and active users of one or several WITHINGS devices, who agreed to receive notifications from Withings Clinical Operations department, and who have previously acquired a WITHINGS device. They will receive a notification through their WITHINGS application, offering them the opportunity to participate in the study. In case of a positive answer, the user will be redirected to the study information sheet.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prediction of uncontrolled hypertension | 2 years
  Correlation between uncontrolled hypertension, Withings data, and survey answers

SECONDARY OUTCOMES:
Correlation between Framingham risk score and EQ-5D-5L answers and Withings data | 2 years
  Correlation between Framingham risk score and EQ-5D-5L answers and Withings data
Number of Questionnaires answers per participant | 2 years
  Number of Questionnaires answers per participant

CONTACTS AND LOCATIONS:
Overall Officials: de Havenon, MD, Principal Investigator — Yale University School of Medicine, Dept of Neurology
Locations (1):
- Yale University Medical School, Department of Neurology, New Haven, Connecticut, United States